CLINICAL TRIAL: NCT06210867
Title: Factors Associated With Occluding the Upper Esophagus by Paratracheal Force
Status: Not yet recruiting | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Other Study IDs: 10-2022-111
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Intubation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aim to identify anatomical factors that affect upper esophageal occlusion during the application of paratracheal pressure.

DETAILED DESCRIPTION:
Measure the sternomental distance, thyromental distance, neck length, neck circumference, Mallampati score, BMI, Neck motion, inter-incisor gap, thyrosternal distance. And analysis these factors are associated with upper esophageal occlusion or not.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 19 years old
* schedule for general anesthesia

Exclusion Criteria:

* Limited neck extension
* Abnormality or anomaly, history of surgery in the neck, esophagus, face, upper airway part.
* Who has weak teeth
* Who has pulmonary aspiration risk

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were scheduled for general anesthesia without a risk of difficult intubation or a history of head and neck surgery.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-02-27 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of esophageal occlusion rate | 10 sec
  Esophageal occlusion is defined as passing an esophageal stethoscope

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, MD,PhD, Study Chair — SMG-SNU Boramae Medical Center
Locations (1):
- Jin-Young Hwang, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warner MA, Warner ME, Weber JG. Clinical significance of pulmonary aspiration during the perioperative period. Anesthesiology. 1993 Jan;78(1):56-62. doi: 10.1097/00000542-199301000-00010. PMID 8424572
- [Background] Lienhart A, Auroy Y, Pequignot F, Benhamou D, Warszawski J, Bovet M, Jougla E. Survey of anesthesia-related mortality in France. Anesthesiology. 2006 Dec;105(6):1087-97. doi: 10.1097/00000542-200612000-00008. PMID 17122571
- [Background] Landreau B, Odin I, Nathan N. [Pulmonary aspiration: epidemiology and risk factors]. Ann Fr Anesth Reanim. 2009 Mar;28(3):206-10. doi: 10.1016/j.annfar.2009.01.020. Epub 2009 Mar 21. French. PMID 19304443
- [Background] Van de Putte P, Vernieuwe L, Jerjir A, Verschueren L, Tacken M, Perlas A. When fasted is not empty: a retrospective cohort study of gastric content in fasted surgical patientsdagger. Br J Anaesth. 2017 Mar 1;118(3):363-371. doi: 10.1093/bja/aew435. PMID 28203725
- [Background] Gautier N, Danklou J, Brichant JF, Lopez AM, Vandepitte C, Kuroda MM, Hadzic A, Gautier PE. The effect of force applied to the left paratracheal oesophagus on air entry into the gastric antrum during positive-pressure ventilation using a facemask. Anaesthesia. 2019 Jan;74(1):22-28. doi: 10.1111/anae.14442. Epub 2018 Oct 4. PMID 30288741